Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses

Protocol CR-6395

Version: 3.0

Date: 28 July 2020

Investigational Products: etafilcon A with PVP cosmetic lenses

Key Words: etafilcon A with PVP cosmetic lenses, daily disposable, dispensing, logMAR visual acuity, subjective vision

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| | OF CONTENTS | |
|---|---|---|
| | COL TITLE, NUMBER, VERSION | |
| SPONS | OR NAME AND ADDRESS | 6 |
| MEDIC | AL MONITOR | 6 |
| AUTHO | PRIZED SIGNATURES | 7 |
| CHANC | GE HISTORY | 8 |
| SYNOP | SIS | 9 |
| COMM | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. IN | TRODUCTION AND BACKGROUND | 17 |
| 1.1. | Name and Descriptions of Investigational Products | 17 |
| 1.2. | Intended Use of Investigational Products | 17 |
| 1.3. | Summary of Findings from Nonclinical Studies | 17 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | |
| 1.5.<br>Study | Relevant Literature References and Prior Clinical Data Relevant to Proposed C. 18 | linica |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 18 |
| 2.1. | Objectives | 18 |
| 2.2. | Endpoints | 18 |
| 2.3. | Hypotheses | 19 |
| 3. TA | RGETED STUDY POPULATION | 19 |
| 3.1. | General Characteristics | 19 |
| 3.2. | Inclusion Criteria | 19 |
| 3.3. | Exclusion Criteria | 20 |
| 3.4. | Enrollment Strategy | 21 |
| 4. ST | UDY DESIGN AND RATIONALE | 21 |
| 4.1. | Description of Study Design | 21 |
| 4.2. | Study Design Rationale | 21 |
| 4.3. | Enrollment Target and Study Duration | 22 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | 22 |
| 5.1. | Test Article Allocation | 22 |
| 5.2. | Masking | 22 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 23 |
| 6. ST | UDY INTERVENTION | 23 |
| 6.1. | Identity of Test Articles. | 23 |

| ( | 5.2. | Ancillar | y Supplies/Products | 24 |
|---|---|---|---|---|
| 6 | 5.3. | Adminis | tration of Test Articles | 24 |
| 6 | 5.4. | Packagii | ng and Labeling | 24 |
| 6 | 5.5. | Storage | Conditions | 25 |
| 6 | 5.6. | Collection | on and Storage of Samples | 25 |
| 6 | 5.7. | Account | ability of Test Articles | 25 |
| 7. | STU | JDY EV. | ALUATIONS | 26 |
| 7 | 7.1. | Time an | d Event Schedule | 26 |
| , | 7.2. | Detailed | Study Procedures | 28 |
| | VIS | SIT 1 | | 28 |
| | VIS | SIT 2 | | 33 |
| | VIS | SIT 3 | | 35 |
| | VIS | SIT 4 | | 39 |
| | FIN | IAL EVA | LUATION | 40 |
| , | 7.3. | Unsched | luled Visits | 41 |
| , | 7.4. | Laborato | ory Procedures | 42 |
| 8. | SU | BJECTS | COMPLETION/WITHDRAWAL | 42 |
| 8 | 3.1. | Complet | ion Criteria | 42 |
| 8 | 3.2. | Withdra | wal/Discontinuation from the Study | 42 |
| 9. | PR] | E-STUD | Y AND CONCOMITANT INTERVENTION/MEDICATION | 43 |
| Ģ | 9.1. | Systemic | e Medications | 43 |
| 10. | D | EVIATIO | ONS FROM THE PROTOCOL | 44 |
| 11. | S | TUDY T | ERMINATION | 45 |
| 12. | P | ROCEDU | JRE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 45 |
| 13. | A | DVERSI | E EVENTS | 47 |
| ] | 13.1. | Defini | tions and Classifications | 47 |
| ] | 13.2. | Assess | sing Adverse Events | 49 |
| | 13.2 | 2.1. C | ausality Assessment | 49 |
| | 13.2 | 2.2. S | everity Assessment | 49 |
| ] | 13.3. | Docur | mentation and Follow-Up of Adverse Events | 50 |
| 1 | 13.4. | Repor | ting Adverse Events | 51 |
| | 13.4 | 4.1. R | eporting Adverse Events to Sponsor | 51 |
| | 13.4 | 4.2. R<br>51 | eporting Adverse Events to the Responsible IEC/IRB and Health Autho 2 | rities |

| 1 | 13.4.3 | B. Event of Special Interest | 52 |
|---|---|---|---|
| 13. | 5. | Reporting of Pregnancy | 52 |
| 14. | STA | ATISTICAL METHODS | 53 |
| 14. | 1. | General Considerations. | 53 |
| 14. | 2. | Sample Size Justification | 53 |
| - | mary | The POWER procedure was used to conduct the power analysis for both and secondary endpoint. The total number of subjects needed to test both and secondary hypothesis is 39. Analysis Populations | h the |
| 14. | 4. | Level of Statistical Significance | 54 |
| 14. | 5. | Primary Analysis | 54 |
| 14. | 6. | Secondary Analysis | 54 |
| 14. | 7. | Other Exploratory Analyses | 54 |
| 14. | 8. | Interim Analysis | 55 |
| 14. | 9. | Procedure for Handling Missing Data and Drop-Outs | 55 |
| 14. | 10. | Procedure for Reporting Deviations from Statistical Plan | 55 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 56 |
| 15. | 1. | Electronic Case Report Form/Data Collection | 56 |
| 15. | 2. | Subject Record | 56 |
| 15. | 3 | ClinicalTrials.gov | 57 |
| 16. | DA | TA MANAGEMENT | 57 |
| 16. | 1. | Access to Source Data/Document | 57 |
| 16. | 2. | Confidentiality of Information | 57 |
| 16. | 3. | Data Quality Assurance | 57 |
| 17. | CLI | NICAL MONITORING | 58 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | 58 |
| 18. | 1. | Study-Specific Design Considerations | 58 |
| 18. | 2. | Investigator Responsibility | 58 |
| 18. | 3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 59 |
| 18. | 4. | Informed Consent | 60 |
| 18. | 5. | Privacy of Personal Data | 61 |
| 19. | STU | JDY RECORD RETENTION | 62 |
| 20. | FIN | ANCIAL CONSIDERATIONS | 62 |
| 21. | PUl | BLICATION | 63 |
| 22. | REI | FERENCES | 63 |

| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 64 |
|---|---|
| APPENDIX B: PATIENT INSTRUCTION GUIDE | 73 |
| APPENDIX C: ASIAN EYE CRITERIA ASSESSMENT PROCEDURE | 74 |
| APPENDIX D: HULA HOOP AND COSMETIC LENS FIT ASSESSMENT | 75 |
| APPENDIX E: | 78 |
| Lens Fitting Characteristics | |
| Subject Reported Ocular Symptoms | 86 |
| Front and Back Surface Lens Deposit Grading Procedure | 88 |
| Determination of Distance Spherocylindrical Refractions | 94 |
| Biomicroscopy Scale | 101 |
| Keratometry | 107 |
| Distance and Near Visual Acuity Evaluation | 109 |
| , Distance LogMAR Visual Acuity Measurement Procedure | 114 |
| Patient Reported Outcomes | 118 |
| White Light Lens Surface Wettability | 120 |
| Visual Acuity Chart Luminance and Room Illumination Testing | 122 |
| Appendix F: COVID-19 Risk Mitigation Guidelines (VWI-0081) | 128 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 138 |
| TABLE OF CONTENTS | |
| Figure 1: Study Flowchart | 14 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | 23 |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |
| Table 4: <u>Disallowed</u> systemic medications (less than 6 months of continual use) | |
| Table 5: Historical CLUE Vision Scores- 1-Week Follow-up Evaluation | 53 |

JJVC CONFIDENTIAL

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses

Protocol Number: CR-6395

Version: 3.0

Date: 28 July 2020

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### **MEDICAL MONITOR**

Title: Senior Principal Research Optometrist Address: 7500 Centurion Parkway, Suite 100

Email: mbishop4@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author/Study | | |
|---|---|---|
| Responsible<br>Clinician | See Electronic Signature Report Senior Principal Research Optometrist, Clinical Science, R&D | DATE |
| Clinical Operations<br>Manager | See Electronic Signature Report Clinical Operations Manager, Clinical Operations, R&D | DATE |
| Biostatistician | See Electronic Signature Report Biostatistician III, Clinical Sciences, R&D | DATE |
| Data Management | See Electronic Signature Report Clinical Project Manager, Data and Systems, R&D | DATE |
| Medical Safety<br>Officer | See Electronic Signature Report Medical Safety Officer | DATE |
| Reviewer | See Electronic Signature Report Clinical Fellow, R&D | DATE |

| Approver | See Electronic Signature Report | |
|----------|---------------------------------|------|
| | | DATE |
| | Director, Specialty Growth | |
| | R&D | |

#### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | | Original Protocol | 04 February<br>2020 |
| 2.0 | | Updated control lens, secondary endpoints/hypothesis, statistical analysis plan, and added Medical Safety Officer to list of approvers | 24 April 2020 |
| 3.0 | | Added COVID risk mitigation<br>guidelines as Appendix F, Revised<br>eligible age range, updated Section<br>13.5 regarding pregnancy during the<br>study. Added Step 1.6 | 28 July 2020 |

#### **SYNOPSIS**

| Protocol Title Clinical Evaluation of Daily Disposable Etafilcon A | |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | |
| Trial Registration | This study will be registered on ClinicalTrials.gov based on the following: confirmatory study meets the requirements for registration. |
| Test Article(s) | Investigational Products: etafilcon A with cosmetic pattern |
| Wear and Replacement | Wear Schedule: Daily Wear |
| Schedules | Replacement Schedule: Daily Disposable |
| Objectives | The primary objective of this study is to evaluate high luminance/high contrast visual performance (Logarithm of Minimal Angle of Resolution [logMAR]) of two investigational cosmetic lenses at lens fitting. |
| | Additional assessments will include: • Subjective Vision (CLUE) • Subjective Comfort (CLUE) • Subjective Handling (CLUE) • logMAR objective vision (high luminance/low contrast and low luminance/high contrast) • Mechanical Lens fit • Cosmetic Lens fit/Hula Hoop • Ocular Physiology |
| Study Endpoints | Primary endpoint: LogMAR visual acuity at fitting using ETDRS charts (CTP-2059). |
| | Other observations (descriptively summarized for each lens type) will include: Subjective Vision (CLUE) Subjective Comfort (CLUE) Subjective Handling (CLUE) logMAR objective vision (high luminance/low contrast and low luminance/high contrast) Mechanical Lens fit Cosmetic Lens fit/Hula Hoop Ocular Physiology |

| Study Design | This will be a randomized, double-masked, bilateral, cross-over, 2 treatment by 2 period dispensing study. There will be 4 visits. There will be a 2 to5 day washout period between treatments. Visit 1: Baseline and eligibility, insert treatment #1, logMAR |
|---|---|
| | vision, post-fit questionnaire, lens fit assessment. Dispense treatment #1 for 6 (±1) days |
| | Visit 2: Follow-up on treatment #1: Subjective questionnaire, logMAR vision, lens fit, and physiology assessment. Washout for 2 to 5 days |
| | Visit 3: Insert treatment #2, logMAR vision, post-fit questionnaire, lens fit assessment. Dispense treatment #3 for 6 (±1) days |
| | Visit 4: Follow-up on treatment #2: Subjective questionnaire, logMAR vision, lens fit. Final evaluation. |
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations. |
| Sample Size | Up to 50 subjects will be enrolled with the aim of approximately 40 subjects completing. |
| Study Duration | The study is expected to last up to 2 months. The enrollment period will also be up to 3 months. |
| Anticipated Study We will aim to recruit up to 50 female subjects, ages | |
| Population | (inclusive). Subject must be habitual contact lens wearers |
| | who have purchased and worn cosmetic/circle contact lenses |
| | in the last 6 months. |
| | We will aim for 60% of the subjects to be self-reported as |
| | Asian with Asian eye characteristics |

| DI TITL OLL I | D |
|---|---|
| Eligibility Criteria | Potential subjects must satisfy all of the following criteria to |
| | be enrolled in the study: |
| | 1. The subject must read, understand, and sign the |
| | STATEMENT OF INFORMED CONSENT and |
| | receive a fully executed copy of the form |
| | 2. Females between 18 and 29 (inclusive) years of age at |
| | the time of screening |
| | 3. Appear able and willing to adhere to the instructions |
| | set forth in this clinical protocol (i.e. willing to wear |
| | only the study lenses and not use habitual lenses |
| | during the dispensing periods) |
| | 4. Be a current soft contact lens wearer in both eyes with |
| | a minimum of 6 hours/day and 5 days/week over the |
| | last month by self-report |
| | 5. Be a current wearer of cosmetic/circle lenses in the last |
| | 6 months, by self-report. |
| | _ · |
| | 6. The subject must be willing to be photographed and/or |
| | video-taped |
| | Inclusion Criteria After Baseline |
| | 7. The subject's vertex corrected spherical equivalent |
| | distance refraction must be in the range of -1.00 D |
| | to -6.00 D (inclusive) in each eye |
| | 8. The subject's refractive cylinder must be less than or |
| | equal to 0.75 D (inclusive) in each eye |
| | · |
| | 9. Have spherical best corrected visual acuity of 20/25 or |
| | better in each eye |

Potential subjects who meet any of the following criteria will be excluded from participating in the study: 1. Currently pregnant or lactating 2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease hepatitis, (eg, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion) 3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion) 4. Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.) 5. Any previous history or signs of a contact lens-related corneal inflammatory event (eg, past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear (at the investigators discretion) 6. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment. 7. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician) Exclusion Criteria after Baseline Eligibility after Baseline: 8. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion) 9. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear. Disallowed See section 9.1

Medications/Interventions

| Measurements and Procedures | logMAR visual acuity, PRO questionnaires (comfort, vision, and handling), lens fit assessment, cosmetic lens fit assessment/hula hoop assessment, and safety parameters (slit lamp findings, entrance/exit visual acuity). |
|---|---|
| Microbiology or Other<br>Laboratory Testing | None |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Tears Naturale re-wetting drops, FluStrips fluorescein strips, Bausch & Lomb Sensitive Eyes plus Saline, or alternative products approved by the Sponsor. |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator

PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome
PVP Polyvinylpyrrolidone
QA Quality Assurance
QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Cosmetic contact lenses can have patterns of varying size and opacities. When designing these cosmetic patterns, it is important to test the performance in a dispensing study on a cosmetic lens wearing population.

In the current study, we will collect objective and subjective performance measures of two investigational cosmetic soft contact lenses.

#### 1.1. Name and Descriptions of Investigational Products

This study will include two types of cosmetic contact lenses. The Control lens and the Test lens are both investigational products. Further details about the test articles are found in Section 6 of this protocol.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigational product is to correct vision. The investigational product contains a cosmetic pattern, so it also affects the visual appearance of the eye. During this dispensing study, each lens type will be worn for approximately 1 week with a 2-5-day washout period between the treatments.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding etafilcon A cosmetic contact lenses refer to the latest version of the Investigator's Brochure (Etafilcon A Investigational Limbal Ring Contact Lenses with polyvinylpyrrolidone [PVP]).

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The following risks/adverse events can be associated with wearing soft contact lenses in general:

- The eyes may burn, sting and/or itch.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers and corneal erosion.
- There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photo-phobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.
- Due to the reduction in light transmittance with cosmetically tinted lenses, some patients may experience visual symptoms while wearing the Study Contact Lenses. In addition, some patients may experience reduced peripheral awareness due to the opaque iris pattern.

There is no direct benefit to the subjects for participating in the study, although they will be able to try out investigational cosmetic contact lenses. The information from this study will aid if the further development and assessment of new potential cosmetic contact lenses.

For the most comprehensive clinical information regarding etafilcon A cosmetic contact lenses with PVP refer to the latest version of the Investigator's Brochure (Etafilcon A Investigational Limbal Ring Contact Lenses with PVP).

## 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

There have been no serious or unanticipated adverse events and no loss of best correct VA reported in pervious etafilcon A with PVP cosmetic contact lens clinical studies. There was one significant adverse event in which was a small non-staining white corneal lesion. The site deemed this as not related to the study lenses as it was present prior to enrollment and stable at the final evaluation.

For the most comprehensive clinical information regarding etafilcon A cosmetic contact lenses with PVP refer to the latest version of the Investigator's Brochure (Etafilcon A Investigational Limbal Ring Contact Lenses with PVP).

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

**Primary Objective** 

The primary objective of this study is to evaluate the objective vision Logarithm of Minimal Angle of Resolution (logMAR) under high illuminance/high contrast lighting conditions of the investigational cosmetic study lenses post lens fitting.

#### 2.2. Endpoints

Primary endpoint

Visual Acuity (logMAR)

Multiple assessments of monocular visual acuity will be made during the study, but the measurements made at post lens fitting using high contrast letters in bright illuminance conditions at distance (4 meters) will be the primary endpoint. VA will be assessed using ETDRS Charts. Additionally, visual acuity will be measured using high and low contrast charts in bright illuminance conditions. Visual acuity will also be measured using normal illumination and normal contrast charts, while wearing goggles. See and and in Appendix E for details regarding the collection of visual acuity (logMAR).

#### Other Endpoints

- Subjective Vision measured via. CLUE
- Subjective Comfort measured via. CLUE
- Subjective Handling measured via. CLUE
- high illumination/low contrast visual acuity
- low illumination/high contrast visual acuity
- Mechanical Lens fit
- Cosmetic Lens fit
- Hula Hoop
- Ocular Physiology

CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.<sup>6</sup>

#### 2.3. Hypotheses

#### Primary Hypothesis

1. The proportion of eyes with corrected distance monocular visual acuity 0.176 logMAR or better (ie, Snellen VA 20/30 or better) using the Test lenses under high illumination/high contrast is superior to 90%.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Females aged 18 to 29 years (inclusive) who are habitual soft contact lens wearers and current wearers of circle/cosmetic contact lenses in the last 6 months will be recruited for this clinical study. While patients within the age range will be eligible to enroll, preference should be given to patients aged 18-24 years. Subjects must meet all the inclusion and none of the exclusion criteria listed in Section 3.2.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
- 2. Females between 18 and 29 (inclusive) years of age at the time of screening

- 3. Appear able and willing to adhere to the instructions set forth in this clinical protocol (i.e. willing to wear only the study lenses and not use habitual lenses during the dispensing periods)
- 4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report
- 5. Be a current wearer of cosmetic/circle lenses in the last 6 months, by self-report.
- 6. The subject must be willing to be photographed and/or video-taped

#### Inclusion Criteria after Baseline

- 7. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye
- 8. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye
- 9. Have spherical best corrected visual acuity of 20/25 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

#### Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating
- 2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg, rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion)
- 3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion)
- 4. Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.)
- 5. Any previous history or signs of a contact lens-related corneal inflammatory event (eg, past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear (at the investigators discretion).
- 6. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment
- 7. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician)

#### Exclusion Criteria after Baseline

8. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion)

9. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials by a market research company.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This is a 4-visit, bilateral, dispensing, randomized, double-masked, 2×2 crossover trial. A total of approximately 50 subjects will be enrolled with a target of 40 subjects to complete the study.

The study begins with an initial visit (Visit 1). If a subject is found to meet all eligibility criteria, they will be randomized to one of two lens wear sequences (Test/Control or Control/Test) in a bilateral fashion.

If the subject is dispensed study lenses at the initial visit, three additional visits will be conducted. Subjects will return for their first follow-up visit (Visit 2) approximately 1-week after the initial visit. After Visit 2, subjects will undergo a washout period between 2 to 5 days, where subjects will be instructed to wear their habitual contact lenses. After the washout period subjects will return for Visit 3, where they will be dispensed their second study lens per the randomization schedule. Subjects will return for their first follow-up for visit, their second study lens and final evaluation (Visit 4) approximately 1-week after Visit 3.

Subjects will be advised to wear the study lenses at least six (6) hours per day during the 5-7 day dispensing periods.

#### 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. A 2×2 bilateral crossover design was considered to be the optimal design since the study period is relatively short the design can be cost effective and more efficient comparisons between treatments can be made than compared a parallel study since fewer subjects are required to achieve the same pre-specified statistical power. Each subject will act as their own control to reduce the influence of potential confounding factors such as age, gender and vision correction. A 2 to 5-day washout between study lens wear will be implemented to help reduce any potential bias.

A post hoc meta-analysis including CR-5956<sup>5</sup> may be performed at the discretion of the study responsible clinician and included in the clinical study report of the current study CR-6395.

#### 4.3. Enrollment Target and Study Duration

Approximately 50 female ages 18 to 29 years (inclusive) who are habitual soft contact lens wearers and who have purchased and worn circle/cosmetic contact lenses in the last 3 months, will be enrolled in this 4-visit, multi-site clinical study. We will aim to have approximately 60% of the enrolled subjects of Asian descent and with Asian eye characteristics (Appendix C). Additionally, we will aim to enroll subjects who are more frequent beauty contact lens wearers (at least once a month for the last 6 months).

Subjects may be screened over the telephone and invited to the site for screening and enrollment procedures. Enrollment is defined as execution of the informed consent and/or assent form.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×2 crossover design. A computer-generated randomization scheme will be used to randomly assign subjects, in block of 2, to one of the two possible lens wear sequences: Test/Control or Control/Test. The random scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment per the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- O Subject meets all the inclusion / exclusion criteria
- o Subject history and baseline information has been collected.

#### 5.2. Masking

The subjects and the investigators will be masked. Both the test and control lens will have the same cosmetic pattern.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The Clinical Supply Unit will generate a unique code for all study lenses. The investigational lenses will have nearly identical labels, differing only in the product specifications and lens code, to maintain masking. Subjects will be dispensed lenses by the lens code in accordance with the randomization scheme provided by the study statistician.

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme.
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Control | Test |
|---|---|---|
| Name | Etafilcon A with PVP with | Etafilcon A with PVP with |
| | cosmetic pattern- Green0 Pilot | cosmetic pattern Green- Line |
| | Line | 26 |
| Manufacturer | Johnson & Johnson | Johnson & Johnson |
| Lens Material | Etafilcon A | Etafilcon A |
| Nominal Base Curve @ | 8.5 mm | 8.5 mm |
| 22°C | | |
| Nominal Diameter @ | 14.2 mm | 14.2 mm |
| 22°C | | |

| Nominal Distance | -1.00 to -6.00 D | -1.00 to -6.00 D |
|-----------------------|------------------|------------------|
| Powers (D) | | |
| Modality in Current | Daily | Daily |
| Study | | |
| Replacement | Daily | Daily |
| Frequency | | |
| Packaging Form (vial, | Blister | Blister |
| blister, etc.) | | |

Each subject will wear approximately 12 of each lens type.

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Sensitive Eyes Plus (Bausch & Lomb) or country-specific alternative approved by the sponsor, FluStrips (Contacare) or country-specific alternative approved by the sponsor, and Tears Naturale Free (Alcon) or country-specific alternative approved by the sponsor.

Table 2: Ancillary Supplies

| | | Solution | |
|---|---|---|---|
| | Sensitive Eyes | Tears Naturale | FluStrips |
| | plus Saline (or | Free (or other | Fluorescein (or |
| Solution Name/Description | other sponsor- | sponsor- | other sponsor- |
| | approved | approved | approved |
| | product) | product) | product) |
| | Bausch & Lomb | Alcon | Contacare |
| Manufacturer | | | Ophthalmics |
| Manufacturer | | | Diagnostics |
| | | | (EOU) |
| Preservative | None | None | None |
| Other distinguishing items (dye, | NA | NA | D&C Yellow No. |
| packaging, approval status, etc. | | | 8, 0.6 mg |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be over-labeled to mask the subject/Investigators to the identity of the lens. The labels will meet the country-specific labeling guidelines for clinical studies involving investigational contact lenses. The test articles will be in plastic bags as the secondary packaging form.



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

No samples will be collected as part of the study procedures.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will destroy all unused test articles.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately</u>.

Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Washout | Visit 3 | Visit 4 |
|---|---|---|---|---|---|
| | Screening, | Treatment | | Dispense | Treatment |
| | Baseline, | 1 Follow- | | Treatment | 2 Follow- |
| | Dispense | up, | | 2 | up, |
| | Treatment | Washout | | | Final |
| | 1 | | | | Evaluation |
| Time Point | Day 0 | $6\pm1$ | 2 - 5 | 2-5 days | Day $6 \pm 1$ |
| | | days from | days | from V2 | days from |
| | | V1 | | | V3 |
| Estimated Visit Duration | 2 hours | 1 hour | | 1 hour | 1 hour |
| Study Informed Consent | X | | | | |
| Inclusion/Exclusion | X | | | | |
| Screening Criteria | | | | | |
| Demographics | X | | | | |
| Medical History & | X | X | | X | X |
| medication review | | | | | |
| Habitual Lens Info | X | | | | |
| CLUE Baseline | X | | | | |

| Visit Information | Visit 1 | Visit 2 | Washout | Visit 3 | Visit 4 |
|---|---|---|---|---|---|
| | Screening, | Treatment | | Dispense | Treatment |
| | Baseline, | 1 Follow- | | Treatment | 2 Follow- |
| | Dispense | up, | | 2 | up, |
| | Treatment | Washout | | | Final |
| | 1 | | | | Evaluation |
| Time Point | Day 0 | 6 ± 1 | 2 - 5 | 2-5 days | Day 6 ± 1 |
| | | days from | days | from V2 | days from |
| | | V1 | | | V3 |
| Estimated Visit Duration | 2 hours | 1 hour | | 1 hour | 1 hour |
| HVID | X | | | | |
| Keratometry | X | | | | |
| Entrance/Exit VA | X | X | | X | X |
| Subjective Refraction | X | | | | |
| Biomicroscopy | X | X<br>X | | X<br>X | X |
| Subject Reported Ocular | X | X | | X | X |
| Symptoms | | | | | |
| Eligibility after baseline | X | | | | |
| exam | | | | | |
| Randomization | X | | | | |
| Lens Fitting #1 | X | | | | |
| Lens Fitting #2 | | | | X | |
| Over- | X | | | X | |
| refraction/optimization | | | | | |
| CLUE Post-Fit | X | | | X | |
| CLUE Follow-Up | | X | | | X |
| LogMAR VA | X | | | X | |
| Cosmetic Lens Fit | X | X | | X | X |
| Assessment | | | | | |
| Hula Hoop Assessment | X | X | | X | X |
| Lens Fit Assessment | X | X | | $\mathbf{X}$ | X |
| Wettability Characteristics | X | X | | X<br>X | X |
| Lens Surface/Deposits | X | X | | X | X |
| Assessment | | | | | |
| Lens Dispensing & | X | | | X | |
| instruction | | | | | |
| Washout instructions | | X | | | |
| Adverse Event Review | | X | | X | X |
| Final Evaluation | | | | | X |

### 7.2. Detailed Study Procedures

VISIT 1

The subjects must present to Visit 1 wearing their habitual contact lenses.

| | | Visit 1: Screening | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. | |
| 1.2 | Demographics | Record the subject's year of birth, gender, race and ethnicity. | |
| 1.3 | Asian Eye<br>Characteristics | Confirm if the subject meets the criteria listed in Appendix C. | Appendix<br>C |
| 1.4 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. | |
| 1.5 | Habitual Lenses | Questions regarding the subject's habitual lens type, parameters, wear schedule and duration. | |
| 1.6 | Wear time and<br>Comfortable Wear<br>Time with Habitual<br>Lenses | Record the subject's wear time and comfortable wear time with their habitual contact lenses. | |
| 1.7 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Visual Acuity, | |
| | | complete Subject Disposition. Visual Acuity,<br>Refraction and Biomicroscopy forms are not<br>required. | |

| | | Visit 1: Baseline | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.8 | CLUE Baseline<br>Questionnaire | The subject will respond to the PRO Baseline CLUE Questionnaire | Appendix<br>A |
| 1.9 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 1.10 | Remove Habitual<br>Contact Lenses | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. | |
| 1.11 | Iris Color | Record iris color in both eyes (self-reported) | |
| 1.12 | Horizontal visible<br>iris diameter (HVID) | Measure the horizontal visible iris diameter for each eye separately using a pd stick in normal room illumination. Measure from the edge of the iris nasally to the edge of the iris temporally. Record in mm to one decimal place. | |
| 1.13 | Keratometry | Record the keratometry readings OD and OS. | |
| 1.14 | Subjective Sphero-<br>cylindrical<br>Refraction | Complete subjective spherocylindrical refraction and record the resultant distance visual acuity (OD, OS and OU) to the nearest letter. Note: The subjects contact lens powers based on the vertexed (12 mm), spherical equivalent must be between -1.00 and -6.00 D. | |
| 1.15 | Slit Lamp Findings | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any slit lamp findings are Grade 3 or higher, the subject is ineligible to continue. Continue to the Final Evaluation Form and dismiss the subject. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. | |
| 1.16 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions<br>must be answered "yes" and all responses to<br>Exclusion Criteria questions must be | |

| answered "no" for the subject to be |
|-------------------------------------|
| considered eligible. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.17 | Lens Selection | Assign the study lens based on the |
| | | randomization scheme. |
| | | Select the contact lens power based on the |
| | | vertexed (12 mm), spherical equivalent |
| | | subjective refraction. |
| 1.18 | Lens Insertion | The Subject inserts the study lenses. Record |
| | | the time of lens insertion. |
| | | Check for lens damage under the slit lamp |
| | | before proceeding with lens settling. |
| | | Replace damaged lenses if applicable. |
| | | Note: Designated site staff should observe the |
| | | insertion process. If it appears that the subject |
| | | attempts to insert a lens that is "inside-out", |
| | | they should interfere to avoid incorrect |
| | | insertion. |
| | | Note 2: If the lens moves excessively on the |
| | | eye after insertion, ask the subject to remove |
| | | the lens, confirm lens is not inverted (correct |
| | | if it is) and reinsert. |
| 1.19 | Lens Settling | Allow the study lenses to settle for a |
| | | minimum of 5 minutes. |
| 1.20 | Subjective Best | Perform subjective best sphere refraction |
| | Sphere Over | over the study lenses with a phoropter (adopt |
| | Refraction | the maximum plus to maximum visual acuity |
| | | (MPMVA) approach and use the duo-chrome |
| | | test for binocular balancing) and record the |
| | | best corrected distance visual acuity to the |
| | | nearest letter (OD, OS, OU). |
| 1.21 | Lens Power | Adjust the lens power if the subject's best |
| | Modification (if | sphere over-refraction is not plano. |
| | applicable) | For each power modification, repeat steps |
| | | (1.16 to 1.19). |
| 1.55 | | Two power modifications are allowed. |
| 1.22 | Visual Acuity | Record the distance Snellen visual acuity (OD, |
| | | OS, and OU) to the nearest letter with the |
| | | study contact lens correction in place. |
| | | Subjects must read the smallest line until at |
| | | least 50% of the letters are read incorrectly. |

| 1.23 | Distance ETDRS | Per , please confirm | |
|---|---|---|---|
| 1.23 | LogMAR Visual | Per , please confirm room illuminance and chart luminance | |
| | Acuity | acceptable ranges for both high/low contrast | |
| | | visual acuity testing. | |
| | | 1. Under high illumination and high chart luminance, record the distance (4 meter) ETDRS high contrast visual acuity twice OD (HC1-HC2) and twice OS (HC3-HC4). | |
| | | 2. Under high illumination and high chart luminance, record the distance (4 meter) ETDRS low contrast visual acuity twice OD (LC1-LC2) and twice OS (LC3-LC4). | |
| | | 3. With the goggles on, under normal illumination and chart luminance, record the distance (4 meter) ETDRS high contrast visual acuity twice OD (HC5-HC6 and twice OS (HC7-HC8). Allow subject to adjust to dim condition for 3 minutes. | |
| | | Letter-by-letter results will be recorded into<br>the electronic data capture form, which will<br>calculate the visual performance score for<br>each chart read. | |
| 1.24 | Subject Reported | Subjects will respond to a verbal open-ended | |
| 1.25 | Ocular Symptoms CLUE Post-Fit | symptoms questionnaire. | |
| 1.23 | Questionnaire | The subject will respond to the CLUE Post-<br>Fit Questionnaire | Appendix<br>A |
| 1.26 | Cosmetic Lens Fit | The Cosmetic Lens Assessment will be | Appendix |
| | Assessment (without | assessed by the investigator (without slit- | D |
| | slit-lamp) | lamp) in primary gaze and extreme gaze | |
| | | (right, left, and upgaze) at a normal | |
| | | conversation distance (approximately three (3) feet away from the subject). | |
| 1.27 | Hula Hoop | If there is an unacceptable cosmetic fit in any | Appendix |
| 1.27 | Assessment (without | gaze, the Hula Hoop Assessment will be | D |
| | slit-lamp) | assessed by the investigator (without slit- | |
| | *If unacceptable | lamp) in primary gaze and extreme gaze | |
| | cosmetic fit in any | (right, left, and upgaze) at a normal | |
| | gaze.* | conversation distance (approximately three | |
| | | (3) feet away from the subject). | |

| 1.28 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. |
|---|---|---|
| | | An unacceptable fit is deemed by one of the following criteria: • Presence of limbal exposure (appearance of clear cornea) in any gaze; • Presence of edge lift; • Presence of unacceptable movement (excessive or insufficient) in all three of the following conditions: primary gaze, up gaze, and tightness on push up. |
| | | Note: if lens fit is unacceptable subject will be discontinued from the study. |
| 1.29 | Wettability<br>Characteristics | Record the white light lens wettability of both lenses. |
| 1.30 | Surface Deposits | Record any front and back surface lens deposits. |
| 1.31 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity is 20/30 or better OD and OS • The lens fit is acceptable OD and OS • Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 1.32 | Dispense | <ul> <li>The lenses will be dispensed for a 5 to 7 day wearing period. During this time, they are required to wear the lenses at least 6 hours per day.</li> <li>Dispense enough lenses to last the subject to their scheduled follow-up visit. Do not dispense extras*.</li> <li>The lenses will be worn as daily wear/daily disposable only.</li> <li>Rewetting drops are permitted if needed.</li> </ul> |

| <ul> <li>A patient instruction booklet will be provided.</li> <li>Subjects will be scheduled for their 5-7-day follow-up visit, ensuring that they wear the study lens at least 6 hours on the day of the follow-up visit.</li> </ul> |
|---|
| * Note: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |

#### VISIT 2

The subjects must present to Visit 2 wearing test article for at least six (6) hours on the day of the visit.

| | Visit 2: Treatment 1 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| 2.1. | Adverse Events and | Review the subject's concomitant |
| | Concomitant | medications and record any changes from the |
| | Medications Review | previous study visit. |
| | | Record any adverse events or medical |
| | | history changes from the previous study |
| | | visit. |
| 2.2. | Wearing Time | Record the average wearing time and |
| | | comfortable wearing time. |
| 2.3. | Compliance | Confirm compliance with the prescribed |
| | | wear schedule. |
| 2.4. | J 1 | Subjects will respond to a verbal open-ended |
| | Ocular Symptoms | symptoms questionnaire. |
| 2.5. | CLUE Follow-Up | The subject will respond to the CLUE |
| | Questionnaire | Follow-Up Questionnaire |
| 2.6. | Entrance Visual | Record the distance Snellen visual acuity |
| | Acuity | (OD, OS, and OU) to the nearest letter with |
| | | study contact lens in place. Subjects must |

| | | read the smallest line until at least 50% of the letters are read incorrectly. | |
|---|---|---|---|
| 2.7. | Cosmetic Lens Fit<br>Assessment<br>(without slit-lamp) | The Cosmetic Lens Assessment will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). | Appendix<br>D |
| 2.8. | Hula Hoop Assessment (without slit-lamp) *If unacceptable cosmetic fit in any gaze.* | If there is an unacceptable cosmetic fit in any gaze, the Hula Hoop Assessment will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). | Appendix<br>D |
| 2.9. | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: • Presence of limbal exposure (appearance of clear cornea) in any gaze; • Presence of edge lift; • Presence of unacceptable movement (excessive or insufficient) in all three of the following conditions: primary gaze, up gaze, and tightness on push up. Note: if lens fit is unacceptable subject will be discontinued from the study. | |
| 2.10 | Wettability Characteristics | Record the white light lens wettability of both lenses. | |
| 2.11 | | Record any front and back surface lens | |
| | | deposits. | |
| | Remove lenses | The lenses will be removed and discarded. | |
| 2.13 | Slit Lamp Findings | FDA Slit Lamp Classification Scale will be used to grade the findings. Adverse events shall be documented and followed for significant slit lamp findings. | |

| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
|---|---|---|
| 2.14 | Washout<br>instructions | Subjects are instructed to wear their spectacles or habitual contact lenses for 2-5 days. |
| 2.15 | Exit Visual Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual spectacles (where applicable). Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |

VISIT 3

The subjects must present to Visit 3 not wearing their habitual contact lenses.

| Visit 3: Treatment 2 Treatment | | |
|---|---|---|
| Step | Procedure | Details |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 3.2. | Visual Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with the habitual spectacle correction (if needed) in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 3.3. | Slit Lamp Findings | FDA Slit Lamp Classification Scale will be used to grade the findings. Adverse events shall be documented and followed for significant slit lamp findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 3.4. | Continuance | Confirm the subject is able to continue in the study. |
| 3.5. | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on the vertexed (12 mm), spherical equivalent subjective refraction. |
| 3.6. | Lens Insertion | The Subject inserts the study lenses. Record the time of lens insertion. |

| | | | I |
|---|---|---|---|
| | | Check for lens damage under the slit lamp | |
| | | before proceeding with lens settling. | |
| | | Replace damaged lenses if applicable. | |
| 3.7. | Lens Settling | Allow the study lenses to settle for a | |
| | | minimum of 5 minutes. | |
| 3.8. | Subjective Best | Perform subjective best sphere refraction | |
| | Sphere Over | over the study lenses with a phoropter (adopt | |
| | Refraction | the maximum plus to maximum visual acuity | |
| | | (MPMVA) approach and use the duo- | |
| | | chrome test for binocular balancing) and | |
| | | record the best corrected <u>distance</u> visual | |
| | | acuity to the nearest letter (OD, OS, OU). | |
| 3.9. | Lens Power | Adjust the lens power if the subject's best | |
| | Modification (if | sphere over-refraction is not plano. | |
| | applicable) | For each power modification, repeat steps | |
| | | (3.13-3.16). | |
| | | Two power modifications are allowed. | |
| 3.10 | Visual Acuity | Record the distance Snellen visual acuity | |
| | | (OD, OS, and OU) to the nearest letter with | |
| | | the study contact lens correction in place. | |
| | | Subjects must read the smallest line until at | |
| | | least 50% of the letters are read incorrectly. | |
| 3.11 | Distance ETDRS | Per please confirm | |
| | LogMAR Visual | room illuminance and chart luminance | |
| | Acuity | acceptable ranges for both high/low contrast | |
| | | visual acuity testing. | |
| | | 4. Under high illumination and high chart | |
| | | luminance, record the distance (4 | |
| | | meter) ETDRS high contrast visual | |
| | | acuity twice OD (HC1-HC2) and twice | |
| | | OS (HC3-HC4). | |
| | | 5. Under high illumination and high chart | |
| | | luminance, record the distance (4 | |
| | | meter) ETDRS low contrast visual | |
| | | acuity twice OD (LC1-LC2) and twice | |
| | | OS (LC3-LC4). | |
| | | , | |
| | | 6. With the goggles on, under normal | |
| | | illumination and chart luminance, | |
| | | record the distance (4 meter) ETDRS | |
| | | high contrast visual acuity twice OD | |
| | | (HC5-HC6 and twice OS (HC7-HC8). | |
| | | Allow subject to adjust to dim | |
| | | condition for 3 minutes. | |
| | | T 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
|---|---|---|---|
| | | Letter-by-letter results will be recorded into | |
| | | the electronic data capture form, which will | |
| | | calculate the visual performance score for | |
| | | each chart read. | |
| 3.12 | Subject Reported | Subjects will respond to a verbal open-ended | |
| | Ocular Symptoms | symptoms questionnaire. | |
| 3.13 | CLUE Post-Fit | The subject will respond to the CLUE Post- | |
| | Questionnaire | Fit Questionnaire | Appendix |
| | | | A |
| 3.14 | Cosmetic Lens Fit | The Cosmetic Lens Assessment will be | Appendix |
| | Assessment | assessed by the investigator (without slit- | D |
| | (without slit-lamp) | lamp) in primary gaze and extreme gaze | |
| | | (right, left, and upgaze) at a normal | |
| | | conversation distance (approximately three | |
| | | (3) feet away from the subject). | |
| 3.15 | Hula Hoop | If there is an unacceptable cosmetic fit in any | Appendix |
| | Assessment | gaze, the Hula Hoop Assessment will be | D |
| | (without slit-lamp) | assessed by the investigator (without slit- | |
| | *If unacceptable | lamp) in primary gaze and extreme gaze | |
| | cosmetic fit in any | (right, left, and upgaze) at a normal | |
| | gaze.* | conversation distance (approximately three | |
| | | (3) feet away from the subject). | |
| 3.16 | Subjective Lens Fit | Evaluate overall lens fit acceptance | |
| | Assessment | (acceptable or unacceptable) based on | |
| | | centration, movement and other fitting | |
| | | characteristics. | |
| | | An unacceptable fit is deemed by one of the | |
| | | following criteria: | |
| | | Presence of limbal exposure | |
| | | (appearance of clear cornea) in any | |
| | | gaze; | |
| | | Presence of edge lift; | |
| | | <ul> <li>Presence of unacceptable movement</li> </ul> | |
| | | (excessive or insufficient) in all three of | |
| | | the following conditions: primary gaze, | |
| | | up gaze, and tightness on push up. | |
| | | ap 5020, and agranous on paon ap. | |
| | | Note: if lens fit is unacceptable subject will | |
| | | be discontinued from the study. | |
| 3.17 | Wettability | Record the white light lens wettability of | |
| | Characteristics | both lenses. | |
| 3.18 | Surface Deposits | Record any front and back surface lens | |
| | • | deposits. | |

| 3.19 | Continuance | <ul> <li>For the subject to continue in the study, they must meet all three of the following criteria:</li> <li>Visual acuity is 20/30 or better OD and OS</li> <li>The lens fit is acceptable OD and OS</li> <li>Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject.</li> <li>Subject is willing to wear the lenses for the dispensing period for 6 hours per day and will not wear their habitual lenses during the dispensing period.</li> </ul> |
|---|---|---|
| 3.20 | Dispense | The lenses will be dispensed for a 5 to 7 day wearing period. During this time, they are required to wear the lenses at least 6 hours per day. • Dispense enough lenses to last the subject to their scheduled follow-up visit. Do not dispense extras*. • The lenses will be worn as daily wear/daily disposable only. • Rewetting drops are permitted if needed. • Subjects will be scheduled for their 1-week follow-up visit, ensuring that they wear the study lens at least 6 hours on the day of the follow-up visit. * Note: In the event a lens is lost or damaged, the subject will return to the |
| | | clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |

# VISIT 4

The subjects must present to Visit 4 wearing test article for at least six (6) hours on the day of the visit.

| the visit. | Visit 4: Treatment 2 Follow-Up | | |
|---|---|---|---|
| Step | ep Procedure Details | | |
| 4.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. | |
| | | Record any adverse events or medical history changes from the previous study visit. | |
| 4.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | |
| 4.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 4.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 4.5. | CLUE Follow-Up<br>Questionnaire | The subject will respond to the CLUE Follow-Up Questionnaire | |
| 4.6. | Preference questions | The subject will respond to the preference Follow-Up Questionnaire | |
| 4.7. | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with study contact lens in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 4.8. | Cosmetic Lens Fit<br>Assessment<br>(without slit-lamp) | The Cosmetic Lens Assessment will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). | Appendix<br>D |
| 4.9. | Hula Hoop<br>Assessment<br>(without slit-lamp)<br>*If unacceptable<br>cosmetic fit in any<br>gaze.* | If there is an unacceptable cosmetic fit in any gaze, the Hula Hoop Assessment will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). | Appendix<br>D |
| 4.10 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |

| | | An unacceptable fit is deemed by one of the following criteria: • Presence of limbal exposure (appearance of clear cornea) in any gaze; • Presence of edge lift; • Presence of unacceptable movement (excessive or insufficient) in all three of the following conditions: primary gaze, up gaze, and tightness on push up. Note: if lens fit is unacceptable subject will be discontinued from the study. |
|---|---|---|
| 4.11 | Wettability | Record the white light lens wettability of |
| | Characteristics | both lenses. |
| 4.12 | Surface Deposits | Record any front and back surface lens |
| | | deposits. |
| 4.13 | Remove lenses | The lenses will be removed and discarded |

# FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study |
| | | successfully. If subject discontinued from the |
| | | study, indicate the reason. |
| F.2 | Exit Slit Lamp | FDA Slit Lamp Classification Scale will be |
| | Biomicroscopy | used to grade the findings. If no slit lamp |
| | | finding is noted on the EDC form it is |
| | | considered as a zero "0" Grade for all |
| | | observations listed. |
| | | After the slit lamp examination, at the |
| | | discretion of the Investigator, rinse the |
| | | subject's eyes thoroughly with preservative- |
| | | free saline. |
| F.3 | Exit Visual Acuity | Record the distance Snellen visual acuity |
| | | (OD, OS, and OU) to the nearest letter with |
| | | their habitual spectacles (where applicable). |
| | | Subjects must read the smallest line until at |
| | | least 50% of the letters are read incorrectly. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject. If subjects only require dispensing of test article, additional testing is not required.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit as appropriate.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |
| U.4 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS, and OU). (as appropriate) |

| Unscheduled Visit | | |
|---|---|---|
| Step | Procedure | Details |
| U.5 | Slit Lamp | FDA Slit Lamp Classification Scale will be |
| | Biomicroscopy | used to grade the findings. If the clearance of |
| | | the fluorescein needs to be expedited, |
| | | preservative-free rewetting drops may be |
| | | instilled. |
| U.6 | Dispensing | Additional lenses may be dispensed. |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual |
| | | acuity (OD, OS, and OU) to the nearest letter. |

## 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent and/or assent;
- they are eligible;
- Completed all study visits;
  - Have not withdrawn/discontinued from the study for any reason described in Section 8.2

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent and/or assent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (eg the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity, as appropriate.

- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow-up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: See section 9.1 Concomitant therapies that are disallowed include: See section 9.1

## 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film. A summary of disallowed medications is shown in Table 4. Subjects taking these medications on a continual, routine basis that have demonstrated successful contact lens wear for at least 6 months will generally be allowed to participate in this study. Subjects taking these medications on a routine basis but for less than 6 months will not be allowed to participate in the study.

NOTE: That subjects taking these medications on a temporary basis (e.g., antihistamines for seasonal allergy) will be allowed to participate if the medication has sufficient time to leave the body prior to the study. This is dependent on the half-life of the drug, body weight / fat, age, genetics, liver / kidney function, and metabolism of the subject. Given these unknowns, subjects taking the medications on a temporary basis must have ceased that medication at least 2 weeks prior to signing the informed consent.

Table 4: Disallowed systemic medications (less than 6 months of continual use).

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Estrogens* | Menopause, osteoporosis, vaginitis | Vagifem, Estrace, Climara, Vivelle-Dot, Premarin, Minivelle, etc., |
| Antihistamines** | Allergic rhinitis, sedation, hives, allergic conjunctivitis, skin allergy, itching, motion sickness | Hydroxyzine, Promethagan,<br>Phenadoz, Vistaril, Claritin,<br>Zyrtec, Astepro, Astelin, Optivar,<br>Pataday, Allegra, Benedryl, etc.,<br> |

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Anticholinergics | Irritable bowel syndrome,<br>Parkinson's disease, peptic ulcer,<br>cystitis, nasal congestion, cold<br>symptoms, overactive bladder,<br>COPD | Symax SL, Homax SL, Cogentin, |
| Beta-blockers | Hypertension, angina, heart attack, migraine, artrial fibrillation, andrenal cancer, essential tumor, glaucoma | 1 , 1 , |
| Psychotropies | Antipsychotic (schizophrenia, mania), antidepression, antiobsessive, antianxiety, mood stabilizer, stimulants (ADHD) | Zoloft, Celexa, Prozac, Lexapro,<br>Effexor, Cymbalta, Ativan,<br>Xanax, Desyrel, Wellbutrin, etc.,<br> |
| Vitamin A<br>analogs | Cystic acne | Isotretinoin |

<sup>\*</sup>Contraceptive medication not included in this category

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation".

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature. The informed consent must also not be contradicted by the deviation.

Protocol waivers are prohibited.

<sup>\*\*</sup>Antihistamines allowed if taken continuously and demonstrated successful wear while taking the medication, or if they stopped taking the medication for at least 2 weeks prior to enrollment

For the dispensing period (following visit 1 and visit 3), if the subject only wears the study lenses for 4 or 8 days it would be a minor deviation. If the subject wears the lenses for 3 or less or 9 or more days it would be a major deviation.

For the washout period (between visit 2 and visits 3), if the duration is 1 or less or 10 or more days it would be a major deviation.

For the study lens wear time on the day of visit 2 and visit 4, if the subject presents having worn the study lenses 2-5 hours it would be a minor deviation. If the subject presents having worn the study lenses 1 hour or less it would be a major deviation.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

• Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."

- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (Refer to Form for test article return instructions).

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect

Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

**NOTE 1:** to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

**NOTE 2** to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."<sup>1</sup>

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article,

if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2).
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown.
- Actions Taken none; temporarily discontinued; permanently discontinued; other.

# 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

## 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

# 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if related to the visual system.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the

infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

## 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

# **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

• Notify the Sponsor immediately.

- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

Not applicable

#### 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes.

Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

## 14.1. General Considerations

Statistical analysis will be undertaken by the study biostatistician. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables, and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

# 14.2. Sample Size Justification

Approximately 50 eligible subjects will be enrolled to target approximately 40 subjects to complete the study. The sample size was calculated to test both the primary hypothesis with a 2-sided type I error of 5% and a minimum of power of 80%.

Based on historical data from where the same Test lens was utilized, the proportion of eye at lens fitting for distance monocular high luminance high contrast was 0.995 and the correlation between the left and right eyes was 0.627. Using this information the total number of subjects needed to achieve the primary hypothesis is 34 subjects. To account for subject dropout this study will target to enroll approximately 50 subjects with the aim to complete approximately 40 subjects.

14.3. The POWER procedure was used to conduct the power analysis for both the primary and secondary endpoint. The total number of subjects needed to test both the primary and secondary hypothesis is 39. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

#### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

#### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

## 14.5. Primary Analysis

## Visual Acuity (logMAR)

Distance monocular high luminance high contrast visual acuity data will be dichotomized into two groups where Y=1 if subjects VA is below 0.176 logMAR and Y=0 otherwise; Y will be analyzed using a generalized linear mixed model with the logit as the link function. Sequence of lens wear, study period and lens type will be included in the model as fixed effects. Other characteristics such as age may be included as covariates in the model. Site will be included as a random effect (G-side). The covariance between residual errors from the same subject and eye across study periods will be modeled using either homogenous compound symmetry (CS) or unstructured (UN). The structure that returns the lowest finite-sample corrected Akaike's Information criterion<sup>7</sup> will be selected as the structure that best fits the model. The Kenward and Roger method,<sup>8</sup> will be used for the denominator degrees of freedom. The proportion of eye with 0.176 logMAR or better while wearing the Test lens will be estimated using a 95% confidence interval for the estimated proportion.

The null and alternative hypothesis to test for superiority of the Test relative to the pre-defined threshold 0.176 logMAR is as follows:

$$H_o: P_{Test} \le 90\%$$
  
 $H_A: P_{Test} > 90\%$ 

Superiority will be declared if the lower limit of the 95% confidence for the estimated proportion of eyes with distance monocular high luminance high contrast VA better than 0.176 logMAR while wearing the Test lens is above 90%. i.e.  $P(p_{Test} > 90\%) \ge 0.975$ .

### 14.6. Secondary Analysis

Not applicable.

## 14.7. Other Exploratory Analyses

Further statistical exploratory analysis can be undertaken, if necessary, at the discretion of the clinical project leader.

Methods for CLUE will follow the analysis described below:

## **CLUE Scores**

CLUE scores will be analyzed separately by domain using a linear mixed model adjusting for baseline values as a covariate. Sequence of lens wear, study period and lens type. Other characteristics such as race, gender and age may be included in the model as covariates. Site will be included as a random effect (G-side). The covariance between residual errors from the

same subject across study periods will be modeled using either homogenous compound symmetry (CS) or unstructured (UN). The structure that returns the lowest finite-sample corrected Akaike's Information criterion<sup>7</sup> will be selected as the structure that best fits the model. The Kenward and Roger method,<sup>8</sup> will be used for the denominator degrees of freedom.

Comparisons between the Test and Control will be carried out using 2-sided 95% confidence intervals constructed for the least-square means (Test minus Control) at the 1-week follow-up evaluation. The null and alternative hypothesis for CLUE vision scores to test for non-inferiority of the Test lens relative to the Control lens is as follows:

$$H_o$$
:  $\mu_{Test} - \mu_{Control} \le -5$   
 $H_A$ :  $\mu_{Test} - \mu_{Control} > -5$ 

Non-inferiority will be declared if the lower limit of the 95% confidence interval for the least-square mean difference is greater than -5. i.e.  $P(\mu_{Test} - \mu_{Control} > -5) \ge 0.975$ .

### 14.8. Interim Analysis

An interim analysis will be conducted after 20 patients have completed the study, in order to monitor the safety and efficacy of the study lenses. Only descriptive statistics will be provided to the study responsible clinician and the project lead. No statistical analyses will be performed during the interim read. No stopping rules will be applied.

## 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 15 imputations.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

# 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica Express 5.5). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Data Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

## 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

## 15.3 ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov based on the following: confirmatory study meets the requirements for registration.

## 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source

data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

Each subject for this study will complete an assent and a parent or legal guardian must give written informed consent according to local requirements after the nature of the study has been fully explained. The assent and consent forms must be signed before performance of any studyrelated activity. The assent and consent forms that are used must be approved by both the Sponsor and by the reviewing IEC/IRB. The assent and informed consent forms should be in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and GCP guidelines, applicable regulatory requirements, and Sponsor policy. Before entry into the study or pre-screening, the Investigator or an authorized member of the clinical site personnel must explain to the potential subject and parent and/or legal guardian the aims, methods, reasonably anticipated benefits, and potential hazards of the study or pre-screening, and any discomfort it may entail. Subjects and parent and/or legal guardian will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject will receive. Finally, they will be told that the Investigator will maintain a subject identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized Sponsor personnel without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the assent and informed consent form, the subject is authorizing such access and agrees to be contacted

after study completion by health authorities and authorized Sponsor personnel for the purpose of obtaining consent for additional safety evaluations if needed.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>9</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

## 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: <a href="https://www.iso.org/standard/45557.html">https://www.iso.org/standard/45557.html</a>
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: <a href="http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: <a href="https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/">https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/</a>
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Bishop, Meredith. Clinical Study Report -Clinical Report "Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses" published on October 19, 2018.
- 6. Wirth RJ, et al. Development of the Contact Lens User Experience: CLUE Scales. *Optom Vis Sci.* 2016;93(8):801-808.
- 7. Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A comparison of two approaches for selecting covariance structures in the analysis of repeated measurements. *Communications in Statistics-Simulation and Computation*. 1998;27:591–604.
- 8. Kenward MG, Roger JH. Small sample inference for fixed effects from restricted maximum likelihood. *Biometrics*. 1997;53:983-997.
- 9. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 10. EU MDR 2017/745

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)






Protocol 6395




5







Confidential








PRO SPECIFICATIO\_\_\_\_\_\_1 Final 2020-01-24 

8
#### APPENDIX B: PATIENT INSTRUCTION GUIDE

Will be provided separately.

#### APPENDIX C: ASIAN EYE CRITERIA ASSESSMENT PROCEDURE

#### GUIDE TO ANATOMICAL DIFFERENCES BETWEEN ASIAN AND CAUCASIAN EYES

#### 1. Palpebral Aperature (PA)



Asian -usually smaller PA (10.2 - 10.5mm)



Non-Asian - larger PA (11.1mm)

2. Horizontal Eyelid Fissure - (HEF)



Asian -usually smaller HEF (25mm)



Non-Asian - larger HEF (26mm)

#### 3. Upper Lid Angle



Asian -usually angled in and down



Non-Asian - usually an arc

#### 4. Lower Lid Angle



Asian -usually flatter



Non-Asian - usually an arc

#### APPENDIX D: HULA HOOP AND COSMETIC LENS FIT ASSESSMENT

The Cosmetic Lens Acceptance will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject).

In this subjective evaluation, the definition of an Acceptable Cosmetic Fit is: The lens centers well on the eye, and does not provide a level of decentration resulting in undesirable cosmetic effect caused by lens displacement. Below is description and illustration of acceptable and unacceptable cosmetic lens fit.

**Primary gaze:** Instruct the subject to look straight ahead. Confirm the subject has proper head and eye alignment (i.e. not tilting head or turning eyes). Direct the instrument stand light or similar light onto the subject's face. Next, the study doctor shall orient themselves so they are at the same height / eye level as the subject. With the subject looking directly at the study doctor or at a fixation target level with the study doctor's eyes, the study doctor will evaluate primary gaze cosmetic fit acceptance. Have the subject **blink naturally**. Observe if the limbal ring covers the iris / limbal area completely during the inter-blink period.

#### Acceptable Cosmetic Lens Fit (Primary Gaze):

If the <u>limbal ring</u> covers the outer iris / limbal area completely during the inter-blink period then this is recorded as an acceptable cosmetic lens fit. Below is an illustration of an acceptable cosmetic fit.



#### **Unacceptable Cosmetic Lens Fit (Primary Gaze):**

If the iris is visible outside of the <u>outer</u> limbal ring print or if the sclera is visible inside of the <u>inner</u> limbal ring print (i.e. sclera is showing through cosmetic effect layer) during the interblink period when the subject is looking in primary gaze then this would be recorded as unacceptable cosmetic fit. If the investigator records an unacceptable cosmetic lens fit acceptance, the investigator will then record the type of the unacceptable cosmetic fit (iris or sclera) and area where it is occurring (inferior, inferior temporal, temporal, etc..). Example: If

an unacceptable cosmetic fit is recorded because of inferior iris exposure, the investigator would record iris / inferior. Below is an illustration of an unacceptable cosmetic fit.

Note: The investigator will only record what they can see without manipulating the eyelids.



**Extreme gaze:** The study doctor shall orient themselves so they are at the same height / eye level as the subject. Instruct the subject to continue to hold their head in a straight ahead position. Direct the instrument stand light or similar light onto the subject's face. Next, the study doctor will ask the subject to move their eyes in three (3) different gazes (right, left, upgaze) and evaluate the cosmetic fit acceptance in each gaze.

Note 1: After the study doctor has asked the subject to look in a particular gaze (right, left, or upgaze) instruct the subject to blink naturally before evaluating cosmetic acceptance in extreme gaze. Observe if the limbal ring covers the iris / limbal area completely during the inter-blink period.

#### Acceptable Cosmetic Lens Fit (Extreme Gaze):

If the limbal ring covers the outer iris / limbal area during the inter-blink completely then this is recorded as an acceptable cosmetic lens fit.

#### **Unacceptable Cosmetic Lens Fit (Extreme Gaze):**

If the iris is visible outside of the <u>outer</u> limbal ring print or if the sclera is visible inside of the <u>inner</u> limbal ring print (i.e. sclera is showing through cosmetic effect layer) during the interblink period when the subject is looking in extreme gaze then this would be recorded as unacceptable cosmetic fit. If the investigator records an unacceptable cosmetic lens fit acceptance, the investigator shall then record the type of the unacceptable cosmetic fit (iris or sclera) and area where it is occurring (inferior, inferior temporal, temporal, etc...). Example: If an unacceptable cosmetic fit is recorded in extreme left gaze because of nasal sclera exposure and temporal iris exposure, the investigator would record sclera / nasal and iris / temporal. Below is an illustration of an unacceptable cosmetic fit in extreme left gaze.

Note 1: The investigator will only record what they can see without manipulating the eyelids.



#### **HULA HOOP EVALUATION:**

Hula hoop is a dynamic evaluation defined as when the subject blinks the amount of lens movement causes the sclera to become more visible (or apparent) inside of the inner limbal ring print. Then, during the inter-blink period, the lens attempts to correctly realign covering the outer iris / limbal area on the subject's eye (or attempts to correctly realign but does not completely center exposing some amount of sclera that is less visible than compared to immediately after the blink). Hula hoop continues to occur with each blink (i.e. more sclera is visible just after the blink and then becomes less or completely absent as the lens settles).

#### APPENDIX E: CLINICAL TECHNICAL PROCEDURES (CTP)

LENS FITTING CHARACTERISTICS
 SUBJECT REPORTED OCULAR SYMPTOMS
 FRONT AND BACK SURFACE LENS DEPOSIT GRADING
 PROCEDURE
 DETERMINATION OF DISTANCE SPHEROCYLINDRICAL
 REFRACTIONS
 BIOMICROSCOPY
 KERATOMETRY
 DISTANCE AND NEAR VISUAL ACUITY EVALUATION
 DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE
 PATIENT REPORTED OUTCOMES
 WHITE LIGHT LENS SURFACE WETTABILITY
 VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION
 TESTING






















FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE









CR-6395, v3.0




DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS

**Determination of Distance Spherocylindrical Refractions** 
















JJVC CONFIDENTIAL



#### Johnson & Johnson Vision Care, Inc.

Title: **Biomicroscopy Scale Document Type:** Work Instruction Revision Number: 9


#### Johnson & Johnson Vision Care, Inc.

Title: **Biomicroscopy Scale Document Type:** Work Instruction **Revision Number: 9** 

#### Johnson & Johnson Vision Care, Inc.

Title: Biomicroscopy Scale

Document Type: Work Instruction

Revision Number: 9




#### Johnson & Johnson Vision Care, Inc.

Title: **Biomicroscopy Scale Document Type:** Work Instruction **Revision Number: 9** 


#### Johnson & Johnson Vision Care, Inc.

Title: Biomicroscopy Scale

Document Type: Work Instruction

Revision Number: 9






DISTANCE AND NEAR VISUAL ACUITY EVALUATION

## Johnson & Johnson Vision Care, Inc.

Distance and Near Visual Acuity Evaluation Title: **Document Type: Clinical Test Procedure** Revision Number: 3


## Johnson & Johnson Vision Care, Inc.

Distance and Near Visual Acuity Evaluation Title: **Document Type: Clinical Test Procedure** Revision Number: 3

## Johnson & Johnson Vision Care, Inc.

Title: Distance and Near Visual Acuity Evaluation

Clinical Test Procedure

Revision Number: 3


## Johnson & Johnson Vision Care, Inc.

Title: Distance and Near Visual Acuity Evaluation

Document Type: Clinical Test Procedure

Revision Number: 3



DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE

## Johnson & Johnson Vision Care, Inc.

Distance LogMAR Visual Acuity Measurement Procedure Title: **Document Type: Clinical Test Procedure Revision Number: 4** 

## Johnson & Johnson Vision Care, Inc.

Title: Distance LogMAR Visual Acuity Measurement Procedure

Document Type: Clinical Test Procedure

Revision Number: 4



## Johnson & Johnson Vision Care, Inc.



| T141 | Johnson & Johnson | vision Care, inc. | | |
|---|---|---|---|---|
| Title: | Patient Reported Outcomes | | | |
| Document Type: | Procedure | D | inian Namban | |
| | | Rev | ision Number: | 2 |
| | - | | | |

WHITE LIGHT LENS SURFACE WETTABILITY

White Light Lens Surface Wettability



VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

| Johnson & Johnson Vision Care, Inc. | | | |
|---|---|---|---|
| Title: | Visual Acuity Chart Luminance and Room Illumination Testing | | |
| <b>Document Type:</b> | Work Instructions | | |
| _ | | Revisio | on Number: 3 |
| _ | | | |

Johnson & Johnson Vision Care, Inc.

| Title: | Visual Acuity Chart Luminance and Room Illumination Testing |
|---|---|
| <b>Document Type:</b> | Work Instructions |
| | Revision Number: 3 |



# Johnson & Johnson Vision Care, Inc. Visual Acuity Chart Luminance and Room Illumination Testing

Title: Visual Acuity Chart Luminance and Room Illumination Testing

Document Type: Work Instructions

Revision Number: 3



## Johnson & Johnson Vision Care, Inc.

| Title: | Visual Acuity Chart Luminance and Room Illumination Testing |
|---|---|
| <b>Document Type:</b> | Work Instructions |
| | Revision Number: 3 |



# Johnson & Johnson Vision Care, Inc.

| Title: | Visual Acuity Chart Luminance and Room Illumination Testing |
|---|---|
| <b>Document Type:</b> | Work Instructions |
| | Revision Number: 3 |



APPENDIX F: COVID-19 RISK MITIGATION GUIDELINES (VWI-0081)

## Johnson & Johnson Vision Care, Inc.



## Johnson & Johnson Vision Care, Inc.



## Johnson & Johnson Vision Care, Inc.



Johnson & Johnson Vision Care, Inc. **Guidelines for COVID-19 Risk Mitigation** Title: **Document Type:** Work Instruction Revision Number: 2

## Johnson & Johnson Vision Care, Inc.

**Guidelines for COVID-19 Risk Mitigation** Title: **Document Type:** Work Instruction Revision Number: 2

## Johnson & Johnson Vision Care, Inc.

Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Work Instruction Revision Number: 2





## Johnson & Johnson Vision Care, Inc.



## Johnson & Johnson Vision Care, Inc.

Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Work Instruction

Revision Number: 2


Johnson & Johnson Vision Care, Inc. **Guidelines for COVID-19 Risk Mitigation** Title: **Document Type:** Work Instruction Revision Number: 2

#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6395 Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses

Version and Date: 3.0 28 July 2020

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,¹ GCP and ICH guidelines,² the Declaration of Helsinki,³ United States (US) Code of Federal Regulations (CFR),⁴ and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH² regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance from JJVCI pertaining to COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct the study in compliance with local, state and governmental guidelines for COVID-19 risk mitigation.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| - | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |